CLINICAL TRIAL: NCT05802875
Title: Building Resilience During the COVID-19 Pandemic: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Building resilience
Record Dates: First submitted 2023-03-21; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-02

CONDITIONS: Healthy; COVID-19; Distress, Emotional
Keywords: Resilience; MRI
MeSH Terms: conditions — COVID-19 | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RASMUS Resilience Training (Experimental): RASMUS is a systematic, behavior-oriented group training in which the following methods are used: mindfulness exercises, exercises in self-compassion/guided meditations, knowledge transfer by means of a teaching talk/lecture, working out the topics in individual and small group work, group exercises, group discussion and exchange, train coping strategies: somatic, cognitive, and emotional levels, independent reflection on what has been learned, homework, weekly protocols, transfer to everyday life, questionnaires on resilience factors, mindfulness, and self-compassion for self-control, linking the course topics with one another.
  Interventions: Behavioral: RASMUS Resilience Training
- Progressive Muscle Relaxation (Active Comparator): As a relaxation method with scientifically proven effects, progressive muscle relaxation aims at the conscious, voluntary tension and relaxation of certain muscle groups, which can bring the body into a state of deep relaxation. The application is not only effective in patients with various diseases, but also in healthy people.
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: RASMUS Resilience Training — RASMUS stands for "Resilience through mindfulness, self-compassion and self-care" and is a German-language 10-week group resilience program with one training unit per week. The main content of the RASMUS is based on seven resilience factors, i.e. acceptance, optimism, taking responsibility, solution orientation, future orientation, role clarity, and network orientation including the aspects of mindfulness, self-compassion, and self-care.
  RASMUS has been tested and certified according to the German Prevention Standard. The Central Prevention Test Center has awarded the seal of approval for the areas of exercise, nutrition, stress management/relaxation, and addictive substance consumption. Accordingly, this training program has been certified as a prevention course that is recognized by the German statutory health insurance companies. Furthermore, RASMUS can and is already offered as a (group) online course.
  Arms: RASMUS Resilience Training
Behavioral: Progressive Muscle Relaxation — Progressive Muscle Relaxation is a representative relaxation technique used in a wide scope of disorders. Developed by the American physician E.Jacobson in the late 1920s, it is based on the finding that anxiety states are usually accompanied by increased muscle tension, while in resting states the muscles are relaxed. By applying this technique, an individual learns how to relax several muscle groups in the body.
  In the context of the current project, PMR is chosen as the active control condition because it is a broadly accepted and easy-to-implement relaxation exercise that can be offered as a (group) online course and does not include specific contents of RASMUS.
  Arms: Progressive Muscle Relaxation

SUMMARY:
This clinical trial is to test the efficacy of a Resilience Training (RASMUS) compared to an active control condition (Progressive Muscle Relaxation, PMR) on resilience, psychological distress, and other clinical variables in a group of people out of the general population with clinically relevant psychological symptoms in the context of the COVID-19 pandemic. In addition, this randomized, controlled, parallel-group study will test the efficacy of RASMUS and PMR in relation to brain structure, function, and metabolite levels. In summary, the main study examines the efficacy of two potentially helpful interventions to improve mental health, whereas the imaging sub-study investigates the potential effects of these interventions on brain volumetry and cortical thickness, on metabolite levels in stress-related brain regions, on brain responses, as well as on functional brain connectivity and communication.

DETAILED DESCRIPTION:
Theoretical framework: The world is experiencing the evolving situation associated with the outbreak of the Corona Virus Disease-2019 (COVID-19), and there is more of need than ever for stress management and self-care. Several studies pointed out, that the COVID-19 pandemic is associated with highly significant levels of psychological distress that in many cases would meet the threshold for clinical relevance. Mental resilience is critical not only to adapt but also to thrive in these unprecedented times. When stress adversity or trauma strike, resilient people still experience anger, grief and pain, but they are able to keep functioning - both physically and psychologically. Resilience is a dynamic process and can potentially be trained.

Objectives: To test the efficacy of a comprehensive training program aimed at increasing resilience (RASMUS) and an active control condition (PMR) in relation to brain structure, function, and metabolite levels.

Methods: 192 people from the general population in Austria who suffer from psychological distress in the context of the COVID-19 pandemic will be randomly assigned to one of two treatment conditions: RASMUS or PMR. The outcome measurements are performed at the beginning, after the intervention (short-term effect) and at the end of the 6-month follow-up (long-term effect). Study assessments will be conducted via telephone and/or video conferencing platforms, and online questionnaires. RASMUS and PMR will be offered as (group-) online courses via video conferencing platforms. In addition, 100 study participants will be recruited for the neuroimaging sub-study (25/ sex/ condition) and will undergo magnetic resonance imaging (MRI) to investigate brain energy metabolism, functional connectivity, and brain responses during functional MRI. MRI will be performed at baseline, after the intervention (short-term effect) and at the end of a 6-month follow-up (long-term effect).

Innovation: While the main study examines the efficacy of two potentially helpful interventions to improve mental health, the current sub-study investigates the potential effects of these interventions on brain volumetry and cortical thickness, on metabolite levels in stress-related brain regions, on brain responses, as well as on functional brain connectivity and communication.

ELIGIBILITY:
Inclusion Criteria:

* GSI-T score (Mini-SCL) ≥63,
* BRS score <3,
* fluent German speakers,
* written informed consent.

Exclusion Criteria:

* Any psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (verified by Mini International Neuropsychiatric Interview [M.I.N.I.] 7.0.2), a history of nicotine or caffeine dependence is acceptable,
* currently engaged in any form of regular psychological therapy offered by psychologists and/or psychiatrists,
* currently engaged in any form of (group) interventions from other disciplines (social work, pedagogy, coaching, alternative therapy etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Total Change Scores on Resilience Scale for Adults (RSA) among Study Completers | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  RSA is a multifactorial resilience questionnaire, which measures key factors contributing to high resilience, namely family support and cohesion, external support systems, and dispositional attitudes and behaviors. The following areas are investigated: perception of self, planned future, social competence, structural style, family cohesion, and social resources. It consists of 33 items which are to answer on the 7-point response scale

SECONDARY OUTCOMES:
Total Change Scores on World Health Organization Quality of Life (WHOQOL BREF) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The WHOQOL BREF (short form) is a tool assessing the subjective quality of life. It is a self-assessment, 24-item instrument widely used in international trials and consists of 4 domains: physical, psychological, social, and environment.
Total Change Scores on Affective Style Questionnaire (ASQ) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The ASQ is a 20-item scale measuring the three affective styles concealing, adjusting, and tolerating, on a 5-point Likert scale ranging from (1) = "not true of me at all" to (5) = "extremely true of me".
Total Change Scores on Self-Compassion Scale (SCS-D) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The SCS-D short form is a questionnaire for assessment of self-compassion which comprises 12 items with six subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. The questions are to be answered on a 5-point Likert scale from 1 = "very rarely" to 5 = "very often".
Total Change Scores on Mindful Attention and Awareness Scale (MAAS) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The MAAS is used to record self-assessed dispositional mindfulness in following three characteristics: (1) intentional, (2) related to the present moment, and (3) non-judgmental. The questionnaire includes 15 self-related statements which should be answered on a 6-point Likert scale ranging from (1) = "almost always" to (6) = "almost never".
Total Change Scores on Perceived Stress Scale (PSS-10) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  With PSS-10 Scale respondents report the degree to which situations in one's life have been unpredictable, uncontrollable, and overloaded in the past month on a 5-point Likert scale ranging from (0) = "never" to (4) = "very often".
Total Change Scores on Brief COPE Inventory (COPE) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  Brief COPE Inventory is applied to assess subjects disposition for using adaptive and maladaptive coping strategies. The maladaptive coping strategies include: denial, substance use, behavioural disengagement, self-distraction, self-blame. The adaptive coping strategies in turn are: active coping, emotional support, expression of emotions, instrumental support, positive reinterpretation, planning, humor, and acceptance.
Total Change Scores on Insomnia Severity Index (ISI) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The ISI is a brief self-report instrument measuring the subjects' perception of insomnia. The ISI comprises seven items assessing the severity of sleep-onset and sleep maintenance difficulties, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a 0 - 4 scale and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
Total Change Scores on The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The ASSIST is used to assess smoking, alcohol and drugs use
Total Change Scores on Brief Symptom Checklist (BSCL) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The BSCL is the extended version of the Mini-SCL and records subjectively perceived impairment of a person through 53 physical and psychological symptoms. It offers a multi-dimensional evaluation with the possibility of repeated measurements. Psychological stress is measured using nine scales: aggressiveness / hostility, anxiety, depression, paranoid thinking, phobic fear, psychoticism, somatization, insecurity in social contact, compulsiveness and three global parameters: Global Severity Index (GSI), Positive Symptom Distress Index (PSDI) and the Positive Symptom Total (PST)
Total Change Scores on Fatigue Assessment Scale (FAS) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The general fatigue questionnaire consists of 10 items in total, five reflecting mental fatigue and physical fatigue. A score of ≥22 is used as a threshold to determine the presence of relevant fatigue.
Total Change Scores on Hospital Anxiety and Depression Scale (HADS) | Baseline (T1), 10 weeks (post treatment) (T2) and 6-months follow-up (T3)
  The HADS consists of two subscales measuring symptoms of depression (7 items) and anxiety (7 items) on a four-point Likert-Scale

OTHER OUTCOMES:
Mini International Neuropsychiatric Interview (M.I.N.I.) | Screening (T1)
  Any DSM-5 psychiatric disorders will be screened with M.I.N.I. 7.0.2 on the recruitment stage. The M.I.N.I. is a validated, structured, diagnostic interview tool with high diagnostic reliability, consisting of questions that parallel symptoms in the Diagnostic and Statistical Manual of Mental Disorders.
The Brief Resilience Scale (BRS) | Screening (T1)
  The BRS measures the ability to recover from stress and is the only scale not simply assessing factors that may favor mental health despite adversities. While most resilience assessments look into the factors that develop resilience, the BRS is a self-rating questionnaire aimed at measuring an individuals' ability to "bounce back from stress". This instrument consists of three positively worded and three negatively worded items that relate to the individual's ability to bounce back from adversity.
Mini Symptom Check List (Mini-SCL) | Screening (T1)
  The Mini-SCL was primarily developed as a sensitive screening instrument and for outcome measurement. It comprises three scales, each with six items from the SCL-90®-S: Depressivity, Anxiety and Somatization as well as a global index (GSI) for recording the psychological stress within the past seven days. T-score of 63 is suggested as a cut-off score to indicate significant distress.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Hofer, Dr., Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project Website — https://www.resilienz-tirol.at/